CLINICAL TRIAL: NCT02204579
Title: Open-label Dose Escalation Study Evaluating the Safety, Tolerability, Pharmacodynamics and Pharmacokinetics of Intravenous NPSP795 in Autosomal Dominant Hypocalcemia Due to Mutations in the Calcium-sensing Receptor Gene: A Drug Repurposing Study
Brief Title: A Study to Determine the Effects of NPSP795 on the Calcium-sensing Receptor in Subjects With Autosomal Dominant Hypocalcemia as Measured by PTH Levels and Blood Calcium Concentrations
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shire (Industry)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAL-C13-001
Record Dates: First submitted 2014-07-28; First posted 2014-07-30 (Estimated); Results first posted 2016-12-21 (Estimated); Last update posted 2021-08-09 (Actual); Status verified 2021-08

CONDITIONS: Autosomal Dominant Hypocalcemia (ADH)
Keywords: Autosomal Dominant Hypocalcemia; Hypocalcemia; ADH; Hypoparathyroidism
MeSH Terms: conditions — Hypercalciuric Hypocalcemia, Familial; Hypocalcemia; Hypoparathyroidism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- NPSP795 (Experimental): intravenous
  Interventions: Drug: NPSP795

INTERVENTIONS:
Drug: NPSP795

SUMMARY:
This is an open-label study looking at the effects of NPSP795 (a selective calcium receptor antagonist) on activating mutations of the Calcium-sensing receptor in patients with Autosomal Dominant Hypocalcemia. Patients with ADH have low blood calcium levels and an inappropriately increased renal calcium excretion, decreased renal phosphate excretion, and hyperphosphatemia. PTH and blood calcium levels will be tested during and after the IV infusion of NPSP795. Concentrations of NPSP795 and length of time of IV infusion will vary depending on measured levels of ionized calcium.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a heterozygous activating mutation of the CaSR gene (ADH); if not previously confirmed, genetic testing will be performed at the screening visit
* At least 18 years of age
* Body mass index (BMI) ≥ 18.5 to < 39 kg/m2

Exclusion Criteria:

* Diseases or conditions that might compromise any major body system or interfere with the pharmacokinetics of NPSP795
* History of treatment with PTH 1-84 or 1-34 within the previous 6 months
* History of hypocalcemia requiring frequent IV calcium infusions
* History of hypocalcemic seizure within the past 3 months
* Blood 25-hydroxy vitamin D level < 25 ng/mL. If subjects have a blood 25-hydroxy vitamin D level < 25 ng/mL at the outpatient screening visit, they will be prescribed vitamin D replacement. Once the 25-hydroxy vitamin D level is > 25 ng/mL, the subject will be eligible to continue on to the treatment phase of the study
* Estimated glomerular filtration rate (GFR) < 25 mL/minute, and/or abnormal hepatic, hematologic, and/or clotting function
* 12 lead resting electrocardiogram (ECG) with clinically significant abnormalities
* Concomitant medications with the potential to interfere with NPSP795 metabolism
* History of thyroid or parathyroid surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2014-07-18 (Actual); Primary Completion 2015-05-04 (Actual); Study Completion 2015-05-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- National Institute of Health (NIH), Bethesda, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- NPSP795: NPSP795 administered Intravenous (IV) infusion for 10 min on Day 1 if certain criteria for ionized calcium and/or blood parathyroid hormone (PTH) were met, an infusion was administered for either 10 min or 3.5 hours on Days 2 & 3, according to a predefined dose escalation scheme. NPSP795 was administered as a 3.5-hour infusion on Day 4, or the participant underwent discharge procedures.
Period: Overall Study
Arm/Group | NPSP795
Started | 7
Participants Started in Pre-Amendment | 2 (Two participants completed treatment in pre-amendment and were re-enrolled in post-amendment.)
Participants Started in Post-Amendment | 5 (Two participants from pre-amendment were re-enrolled with different identification numbers.)
Treated | 5
Completed | 5
Not Completed | 2
Not completed — Screen failures | 2

BASELINE CHARACTERISTICS:
Arm/Group | NPSP795
Number analyzed (Participants) | 5
Age, Continuous [Mean (Standard Deviation); unit: Years] | 39.8 (15.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Treatment Emergent Serious Adverse Events (TESAEs)
Time Frame: From Day 1 up to safety follow-up assessment (upto Day 17 after discharge)
Population: Safety population included all participants who received at least 1 minute of study drug infusion (pre-amendment and post-amendment).
Measure: Number; unit: participants
Arm/Group | NPSP795
Number analyzed (Participants) | 5
participants
  Participants with TEAEs | 3
  Participants with TESAEs | 1

2. Primary Outcome: Number of Participants With Clinically Significant Vital Signs and Electrocardiogram (ECG) Abnormalities
Time Frame: From Day 1 up to safety follow-up assessment (upto Day 17 after discharge)
Population: Safety population included all participants who received at least 1 minute of study drug infusion (both pre-amendment and post-amendment participants).
Measure: Number; unit: participants
Arm/Group | NPSP795
Number analyzed (Participants) | 5
participants | 0

3. Primary Outcome: Number of Participants With Potentially Clinically Important Laboratory Abnormalities
Time Frame: From Day 1 up to safety follow-up assessment (upto Day 17 after discharge)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | NPSP795
Number analyzed (Participants) | 5
participants | 1

4. Primary Outcome: Number of Participants With Clinically Significant Abnormalities Related to Physical Examination
Time Frame: From Day 1 up to safety follow-up assessment (upto Day 17 after discharge)
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | NPSP795
Number analyzed (Participants) | 5
participants | 1

5. Primary Outcome: Change From Baseline in Ionised Calcium
Time Frame: 10 Minute (min) Infusion Time: within 5 min pre-dose; & post-dose 15, 30, 45, 60, 75, 90, 105 min, and 2, 2.5, 3, 3.5, & 4 hour (hr) 3.5 hr Infusion Time: within 5 min pre-dose; & post-dose 15, 30, 45, 60, 75, 90, 105 min, & 2, 2.5, 3, 3.5, 4, 5, and 8 hr
Population: Post-amendment pharmacodynamic (PD) analysis population included all participants who received at least 5 minutes of the study drug infusion and had at least one PD measurement on at least 1 day of infusion. Here, n=number of participants analysed for specified category at the specified time points in each arm respectively.
Measure: Mean (Standard Deviation); unit: millimole/liter (mmol/L)
Arm/Group | NPSP795 on Day 1 (5 mg/10 Minutes) | NPSP795 on Day 2 (15 mg/3.5 Hours) | NPSP795 on Day 3 (30 mg/3.5 Hours) | NPSP795 on Day 4 (30 mg/3.5 Hours) | NPSP795 on Day 4 (50 mg/3.5 Hours)
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 5
millimole/liter (mmol/L)
  Baseline: number analyzed (Participants) | 5 | 5 | 5 | 3 | 2
  Baseline | 0.972 (0.058) | 0.950 (0.054) | 0.986 (0.045) | 0.933 (0.055) | 1.025 (0.078)
  Change at 4 Hours Post dose: number analyzed (Participants) | 5 | 5 | 5 | 3 | 2
  Change at 4 Hours Post dose | -0.016 (0.027) | 0.010 (0.026) | -0.014 (0.023) | -0.030 (0.046) | -0.015 (0.035)
  Change at 8 Hours Post dose: number analyzed (Participants) | 5 | 5 | 5 | 3 | 2
  Change at 8 Hours Post dose | NA (NA) — Data was calculated for 5 mg/10 minutes infusion until hour 4 only. | -0.034 (0.044) | -0.040 (0.060) | -0.033 (0.046) | -0.060 (0.028)

6. Primary Outcome: Change From Baseline in Serum Calcium
Time Frame: 10 Minutes (min) Infusion Time: within 5 min pre-dose; & post-dose 1, 2, 3, 4, 8 12 hours (hr). 3.5 hr Infusion Time: within 5 min pre-dose; & post-dose 1, 2, 3, 4, 8 12 hr.
Population: Post-amendment PD analysis population included all participants who received at least 5 minutes of the study drug infusion and had at least one PD measurement on at least 1 day of infusion. Here, n=number of participants analysed for specified category at the specified time points in each arm respectively.
Measure: Mean (Standard Deviation); unit: millimole/liter (mmol/L)
Arm/Group | NPSP795 on Day 1 (5 mg/10 Minutes) | NPSP795 on Day 2 (15 mg/3.5 Hours) | NPSP795 on Day 3 (30 mg/3.5 Hours) | NPSP795 on Day 4 (30 mg/3.5 Hours) | NPSP795 on Day 4 (50 mg/3.5 Hours)
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 5
millimole/liter (mmol/L)
  Baseline: number analyzed (Participants) | 5 | 5 | 5 | 3 | 2
  Baseline | 1.914 (0.157) | 1.790 (0.125) | 1.852 (0.132) | 1.677 (0.135) | 1.980 (0.184)
  Change at 12 Hours Postdose: number analyzed (Participants) | 5 | 5 | 5 | 3 | 2
  Change at 12 Hours Postdose | -0.114 (0.141) | -0.042 (0.054) | -0.106 (0.079) | -0.040 (0.053) | -0.270 (0.057)

7. Primary Outcome: Change From Baseline in Urinary Calcium
Time Frame: as for outcome 6
Population: PD analysis population included all participants who received at least 5 minutes of the study drug infusion and had at least one PD measurement on at least 1 day of infusion. Here, n=number of participants analysed for specified category at the specified time points in each arm respectively.
Measure: Mean (Standard Deviation); unit: millimole/liter (mmol/L)
Arm/Group | NPSP795 on Day 1 (5 mg/10 Minutes) | NPSP795 on Day 2 (15 mg/3.5 Hours) | NPSP795 on Day 3 (30 mg/3.5 Hours) | NPSP795 on Day 4 (30 mg/3.5 Hours) | NPSP795 on Day 4 (50 mg/3.5 Hours)
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 5
millimole/liter (mmol/L)
  Baseline: number analyzed (Participants) | 5 | 5 | 5 | 3 | 2
  Baseline | 3.302 (2.283) | 3.912 (3.299) | 2.936 (1.750) | 2.537 (1.968) | 2.065 (1.916)
  Change at 12 Hours Postdose: number analyzed (Participants) | 5 | 5 | 5 | 3 | 2
  Change at 12 Hours Postdose | -0.590 (0.861) | -2.162 (2.027) | -1.188 (1.634) | -1.190 (1.460) | -0.755 (1.082)

8. Primary Outcome: Change From Baseline in Serum Parathyroid Hormone (PTH)
Time Frame: 10 Minutes (min) Infusion Time: within 5 min pre-dose; & post-dose 5, 10, 15, 30 min, & 1, 1.5, 2, 2.5, 3, 3.5, 4, 8 hours (hr). 3.5 hr Infusion Time: within 5 min pre-dose; & post-dose 15, 30 min, & 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 5.5 hr
Population: Post amendment PD analysis population included all participants who received at least 5 minutes of the study drug infusion and had at least one PD measurement on at least 1 day of infusion. Here, n=number of participants analysed for specified category at the specified time points in each arm respectively.
Measure: Mean (Standard Deviation); unit: nanogram/liter (ng/L)
Arm/Group | NPSP795 on Day 1 (5 mg/10 Minutes) | NPSP795 on Day 2 (15 mg/3.5 Hours) | NPSP795 on Day 3 (30 mg/3.5 Hours) | NPSP795 on Day 4 (30 mg/3.5 Hours) | NPSP795 on Day 4 (50 mg/3.5 Hours)
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 5
nanogram/liter (ng/L)
  Baseline: number analyzed (Participants) | 5 | 5 | 5 | 3 | 2
  Baseline | 7.32 (2.93) | 9.14 (3.29) | 9.58 (5.32) | 12.80 (8.68) | 7.40 (3.54)
  Change at 5.5 Hours Postdose: number analyzed (Participants) | 5 | 5 | 5 | 3 | 2
  Change at 5.5 Hours Postdose | NA (NA) — Data for 10 minutes infusion was not calculated at 5.5-hours. | 0.84 (0.86) | 1.92 (1.53) | 0.13 (1.50) | 1.75 (0.64)
  Change at 8 Hours Postdose: number analyzed (Participants) | 5 | 5 | 5 | 3 | 2
  Change at 8 Hours Postdose | 0.60 (1.56) | NA (NA) — Data for 3.5-hours infusions was calculated until hour 5.5 only. | NA (NA) — Data for 3.5-hours infusions was calculated until hour 5.5 only. | NA (NA) — Data for 3.5-hours infusions was calculated until hour 5.5 only. | NA (NA) — Data for 3.5-hours infusions was calculated until hour 5.5 only.

9. Secondary Outcome: Area Under the Plasma Concentration Versus Time Curve (AUC[0-t]) of NPSP795
Time Frame: as for outcome 8
Population: Post amendment pharmacokinetic (PK) analysis population included all participants who received at least 5 minutes of the study drug infusion and had at least one PK measurement on at least 1 day of infusion.
Measure: Mean (Standard Deviation); unit: nanogram*hour per millilitre (ng·h/mL)
Arm/Group | NPSP795 on Day 1 (5 mg/10 Minutes) | NPSP795 on Day 2 (15 mg/3.5 Hours) | NPSP795 on Day 3 (30 mg/3.5 Hours) | NPSP795 on Day 4 (30 mg/3.5 Hours) | NPSP795 on Day 4 (50 mg/3.5 Hours)
Number analyzed (Participants) | 5 | 5 | 5 | 3 | 2
nanogram*hour per millilitre (ng·h/mL) | 309.512 (122.601) | 795.766 (294.345) | 1561.746 (546.479) | 1657.057 (650.156) | 2251.818 (568.782)

10. Secondary Outcome: Area Under the Concentration Time Curve Extrapolated to Infinity (AUC0-infinity) of NPSP795
Time Frame: as for outcome 8
Population: Post amendment PK analysis population included all participants who received at least 5 minutes of the study drug infusion and had at least one PK measurement on at least 1 day of infusion.
Measure: Mean (Standard Deviation); unit: nanogram*hour per milliliter(ng·h/mL)
Arm/Group | NPSP795 on Day 1 (5 mg/10 Minutes) | NPSP795 on Day 2 (15 mg/3.5 Hours) | NPSP795 on Day 3 (30 mg/3.5 Hours) | NPSP795 on Day 4 (30 mg/3.5 Hours) | NPSP795 on Day 4 (50 mg/3.5 Hours)
Number analyzed (Participants) | 5 | 5 | 5 | 3 | 2
nanogram*hour per milliliter(ng·h/mL) | 2.672 (1.775) | 5.572 (2.724) | 5.437 (2.587) | 7.648 (3.607) | 4.521 (2.991)

11. Secondary Outcome: Maximum Observed Drug Concentration (Cmax) of NPSP795 in Plasma
Time Frame: as for outcome 8
Population: Post amendment PK analysis population included all randomized participants who received at least 5 minutes of the study drug infusion and had at least one PK measurement on at least one day of infusion.
Measure: Mean (Standard Deviation); unit: nanogram/milliliter (ng/mL)
Arm/Group | NPSP795 on Day 1 (5 mg/10 Minutes) | NPSP795 on Day 2 (15 mg/3.5 Hours) | NPSP795 on Day 3 (30 mg/3.5 Hours) | NPSP795 on Day 4 (30 mg/3.5 Hours) | NPSP795 on Day 4 (50 mg/3.5 Hours)
Number analyzed (Participants) | 5 | 5 | 5 | 3 | 2
nanogram/milliliter (ng/mL) | 301.900 (120.664) | 745.335 (254.205) | 1467.102 (475.343) | 1515.086 (548.056) | 2141.500 (475.706)

12. Secondary Outcome: Elimination Half-life (t1/2) of NPSP795 in Plasma
Time Frame: as for outcome 8
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | NPSP795 on Day 1 (5 mg/10 Minutes) | NPSP795 on Day 2 (15 mg/3.5 Hours) | NPSP795 on Day 3 (30 mg/3.5 Hours) | NPSP795 on Day 4 (30 mg/3.5 Hours) | NPSP795 on Day 4 (50 mg/3.5 Hours)
Number analyzed (Participants) | 5 | 5 | 5 | 3 | 2
hour | 3.013 (0.612) | 3.913 (0.222) | 4.213 (0.449) | 3.839 (0.294) | 4.000 (0.000)

13. Secondary Outcome: Change From Baseline in Fractional Excretion of Calcium (FECa)
Time Frame: 10 Minutes (min) Infusion Time: within 5 min pre-dose; & post-dose 1, 2, 3, 4, 8, 12 hours (hr). 3.5 hr Infusion Time: within 5 min pre-dose; & post-dose 1, 2, 3, 4, 8, 12 hr.
Population: Post-amendment PD analysis population included all participants who received at least 5 minutes of the study drug infusion and had at least one PD measurement on at least 1 day of infusion. Here n=number of participants analysed for specified category at the specified time points in each arm respectively.
Measure: Mean (Standard Deviation); unit: Fraction of excretion
Arm/Group | NPSP795 on Day 1 (5 mg/10 Minutes) | NPSP795 on Day 2 (15 mg/3.5 Hours) | NPSP795 on Day 3 (30 mg/3.5 Hours) | NPSP795 on Day 4 (30 mg/3.5 Hours) | NPSP795 on Day 4 (50 mg/3.5 Hours)
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 5
Fraction of excretion
  FECa: Baseline: number analyzed (Participants) | 5 | 5 | 5 | 3 | 2
  FECa: Baseline | 0.030 (0.023) | 0.031 (0.017) | 0.027 (0.014) | 0.030 (0.011) | 0.026 (0.032)
  FECa: Change at 12 Hours Postdose: number analyzed (Participants) | 5 | 5 | 5 | 3 | 2
  FECa: Change at 12 Hours Postdose | 0.002 (0.005) | 0.002 (0.012) | 0.001 (0.011) | -0.009 (0.018) | 0.002 (0.007)

ADVERSE EVENTS:
Time Frame: From the sign of informed consent form (Day -93) up to safety follow-up assessment (upto Day 17 after discharge)
Arm/Group | NPSP795
Serious Adverse Events (participants affected / at risk) | 1/5
Other Adverse Events (participants affected / at risk) | 3/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NPSP795 (N=5)
Cholelithiasis (Hepatobiliary disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NPSP795 (N=5)
Cholelithiasis (Hepatobiliary disorders) | 1 (1)
Hypersensitivity reaction (Immune system disorders) | 1 (2)
Nipple pain (Reproductive system and breast disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.